CLINICAL TRIAL: NCT04203940
Title: Sutured Versus Cyanoacrylate Glue Mesh Fixation for Inguinal Hernia Repair: A Randomized Controlled Trial
Brief Title: Sutured Versus Cyanoacrylate Glue Mesh Fixation for Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, lecturer of surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Mansoura122
Record Dates: First submitted 2019-12-17; First posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Sutures

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyanoacrylate (Active Comparator): mesh fixation was done using dots of N-butyl 2-cyanoacrylate tissue glue (Histoacryl®).
  Interventions: Procedure: Cyanoacryale
- Suture (Active Comparator): mesh fixation was done with polypropylene 2/0 sutures
  Interventions: Procedure: Suture

INTERVENTIONS:
Procedure: Cyanoacryale — mesh fixation was done using dots of N-butyl 2-cyanoacrylate tissue glue
  Arms: Cyanoacrylate
Procedure: Suture — mesh fixation was done with polypropylene 2/0 sutures
  Arms: Suture

SUMMARY:
Because it avoids direct nerve irritation or entrapment, mesh fixation with tissue adhesive glue seems an optimal option to reduce postoperative pain. Indeed, preliminary results published with different glues all showed promising results with reduced postoperative pain.

This randomized controlled study aimed to compare mesh fixation using N-butyl 2-cyanoacrylate with classical suture fixation in Lichtenstein hernia repair in terms of chronic groin pain, postoperative complications, operative time and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders aging between 18-65 years with primary unilateral uncomplicated inguinal hernia were included.

Exclusion Criteria:

* Patients with bilateral or sliding inguinal hernia.
* incarcerated or strangulated hernia
* recurrent inguinal hernia
* femoral hernia
* patients unwilling to participate in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Pain score at 12 months after surgery | 12 months after hernia repair
  Pain assessed by visual pain scale from 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, M.D., Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided